CLINICAL TRIAL: NCT03197311
Title: A Mobile Application to Monitor Patient's Analgesic Consumption After Minor Oral Surgery.
Brief Title: A Mobile Application for Post-op Analgesic Consumption
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain funding for this research.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-36258
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Tooth Extraction Status Nos; Post Operative Pain; Patient Satisfaction; Narcotic Use; Mobile App
Keywords: Oral surgery; Medication adherence
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app group (Experimental): In addition to receiving standard of care which includes prescription of postoperative narcotic and NSAID analgesics and usual postoperative instructions a customized mobile app will be downloaded to the participant's smartphone to application to monitor postoperative analgesic consumption, disposal and pain control and patient satisfaction for one week after surgery.
  Interventions: Other: Mobile app
- Control group (No Intervention): The control group will receive the standard of care which includes prescription of postoperative narcotic and NSAID analgesics and usual postoperative instructions and a case report form will be used to gather data from the medical record and from a post op telephone survey a week after surgery..

INTERVENTIONS:
Other: Mobile app — A customized mobile application will be developed and downloaded to subjects; smartphones to monitor postoperative analgesic consumption, and disposal; pain control and patient satisfaction. The mobile app will provide notifications for medications and select education links on the prescribed analgesics. Subjects will receive reminders to take medications as directed. Subjects will be able to monitor and report their pain during the first week after surgery.
  Arms: Mobile app group

SUMMARY:
Surgical extraction of third molars is one of the most common outpatient procedures performed by oral surgeons. The prescription of postoperative narcotic and NSAID analgesics is the standard of care practice to relieve symptoms of pain, swelling, and trismus after these procedures. The majority of these patients do not return for follow up unless they experience a problem. There is limited data on whether the patients use the narcotics as directed and what is their practice of disposal of the remaining medications that were not consumed.

In this research the effectiveness of postop analgesic consumption, analgesic disposal practice, pain control, and patient satisfaction will be compared between patients who are randomized to the intervention group who will use a developed mobile application and a control group who will not use the mobile app.

DETAILED DESCRIPTION:
A pilot randomized clinical trial will be conducted to determine if use of a mobile application improves adherence to narcotic analgesic use and their disposal and patient satisfaction post-surgical extraction of third molars in an outpatient setting. Eligible consented subjects will be randomized into either the mobile app group or the control group. Both groups will receive standard of care which includes prescription of postoperative narcotic and NSAID analgesics and usual postoperative instructions.For the mobile group, the Medable Axon Software developed by Stanford University will be used to customize a mobile application that will be used one week post surgery to monitor postoperative analgesic consumption and disposal practices, pain control, and patient satisfaction, In the control group, case report forms will be used to gather data from the electronic medical records and a telephone survey will be done one week post surgery to obtain data on patient satisfaction. A total of 20 consecutive eligible patients will be enrolled in this pilot trial..

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-40 years
* Patients who require two mandibular third molars extracted
* Patients with a smartphone

Exclusion Criteria:

* Patients taking any recreational drugs and medications for chronic pain

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of quantity of postop analgesic (narcotic and non narcotic) medications used. | At the end of 7 days
  Each patient will be given 18-24 tablets the prescription: 1. Acetaminophen with 5mg oxycodone 2. Acetaminophen with 5mg hydrocodone 3. Acetaminophen with 30 mg codine and asked to report each time they take a tablet via the app in the experimental group while the control group will answer the question how many tablets do you have remaining as part of the post survey at the end of 1 week.
Assessment of change in Postoperative pain control | Daily for 7 days post-op (experimental group) and At the end of 7 days (control group)
  The Short Form McGill Pain Questionnaire (SF-MPQ) will be used to assess post-op pain control. It consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. Lower scores are associated with less pain..

SECONDARY OUTCOMES:
Satisfaction with the education received regarding the prescribed medications. | Daily for 7 days post-op (experimental group) and At the end of 7 days (control group)
  Assessment of patient satisfaction using a survey. For the subjects in the experimental group, they will be asked to complete a emoticon survey on the app which would correspond to the following descriptions: Excellent=4, good=3, average=2, poor=1.The subjects in the control group will be asked the same question as part of the post satisfaction survey without the emoticons as a sentence question. A lower score indicates low satisfaction.
Use of the analgesic and post-op care education links on the mobile app. | Daily for 7 days post-op (experimental group) and At the end of 7 days (control group)
  Educational links will be available to view as part of the app and usage will be monitored by website traffic. Higher numbers would indicate greater usage of educational links.

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Chigurupati, DMD, MS, Study Director — Boston University
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No